CLINICAL TRIAL: NCT01120873
Title: Phase 3 Study of 3D in Metabolic Syndrome
Brief Title: The Effect of Metamin 3D on the Lipid and Glucose in Subjects With Metabolic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: I-Te, Lee, Division of Endocrinology and Metabolism, Department of Internal Medicine, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S06203
Record Dates: First submitted 2010-05-05; First posted 2010-05-11 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Metabolic Syndrome
Keywords: Hyperglycemia; dyslipidemia; Hypertension; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Hyperglycemia; Dyslipidemias; Hypertension; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metamin 3D (Experimental): A randomized, double-blinded and placebo-controlled study
  Interventions: Drug: Metamin 3D

INTERVENTIONS:
Drug: Metamin 3D — Metamin 3D is composed by red yeast rice, bitter gourd, chlorella, soy peptide and licorice extract is a commercial product designed by Uni-President enterprises corp in Taiwan
  Other Names: 3D

SUMMARY:
To evaluate the effect of Metamin 3D on improvement of glucose and lipid on Taiwanese subjects with metabolic syndrome.

DETAILED DESCRIPTION:
The Metamin 3D consists of mixed extractives of nature plants, including soy bean protein, bitter melon, red yeast rice, green algae and trisodium glycyrrhizinate. the improvement of lipid and glucose was reported respectively previously. We design a prospective, double-blinded and placebo-controlled study to evaluate the improvement on metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 75 years
* Fasting plasma glucose >= 100 mg/dl
* Triglyceride >= 150 mg/dl
* one of the criteria following

  1. HDL <40 mg/dl in man or <50 mg/dl in woman
  2. Blood pressure >= 135/85 mmHg or anti-hypertension drug treatment
  3. Waist >90cm in man or 80cm in woman
* Signed the inform consent

Exclusion Criteria:

* Fasting plasma glucose > 180mg/dl
* Treated by more than two types oral hypoglycemic agents in past 3 months
* Treated continuously by anti-lipid agents for 3 months in past 6 months
* Treated by thiazolidinedione or digitalis at present
* Serum creatine > 2.5mg/dl
* Liver function (GOT or GPT) more than 3-fold upper limit
* Severe systemic disease by investigator's judgement
* Pregnant or nursing women
* Enrolled in other clinical study in recent 1 month

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Total cholesterol | 12 weeks
  To assess the change of total cholesterol between 0 and 12 weeks

SECONDARY OUTCOMES:
Total cholesterol | 4 and 8 weeks
  To assess the change of lipid profiles during study
Triglycerides | 4 and 8 weeks
  To assess the change of lipid profiles during study
Low-density lipoprotein cholesterol | 4, 8 and 12 weeks
  LDL cholesterol:
  To assess the lipid profiles during study
The plasma insulin by meal tolerant test | 4 and 8 weeks
Glycosylated hemoglobin | 4 and 8 weeks
  HbA1c:
  To assess the glycemic control during the study period
Fasting plasma glucose | 4 and 8 weeks
  withdrawal if fasting glucose greater than 250 mg/dl
Systolic and diastolic blood pressure | 4, 8 and 12 weeks
Triglycerides | 12 weeks
  To assess the change of lipid profiles between 0 and 12 weeks
The plasma glucose by meal tolerant test | 12 weeks
Glycosylated hemoglobin | 12 weeks
  To assess the change of HbA1c between 0 and 12 weeks
Fasting plasma glucose | 12 weeks
  withdrawal if fasting glucose greater than 250 mg/dl
Aspartate aminotransferase | 12 weeks
  GOT:
  To assess the liver functions at 0 and 12 weeks
Alanine aminotransferase | 12 weeks
  GPT:
  To assess the liver functions at 0 and 12 weeks
Creatinine | 12 weeks
  Serum creatinine:
  To assess the renal function at 0 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: I Te Lee, MD, Principal Investigator — Taichung Veterans General Hospital, Taichung
Locations (1):
- Division of Endocrinology and Metabolism, Department of Internal Medicine, Taichung Veterans General Hospital, Taichang, Taiwan

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/entrez/query/static/citmatch.html